CLINICAL TRIAL: NCT00675155
Title: Phase 1 Study to Determine the Efficacy of Using Far Infrared Radiation for Stroke Rehabilitation
Brief Title: Far Infrared Irradiation for Stroke Rehabilitation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-SR-CTP1
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Stroke
Keywords: Apoplexy; Cerebral Stroke; Cerebrovascular Accident; Cerebrovascular Accident, Acute; Cerebrovascular Apoplexy; Cerebrovascular Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Radiation: Far Infrared Radiation (5μm to 20μm wavelength)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Radiation: Far Infrared Radiation (5μm to 20μm wavelength) Far Infrared radiation for 30 to 40 minutes per treatment session.

SUMMARY:
A stroke is a sudden loss of brain function. It is caused by the interruption of flow of blood to the brain (ischemic stroke) or the rupture of blood vessels in the brain (hemorrhagic stroke). This study will investigate the use of far infrared radiation for stroke rehabilitation.

DETAILED DESCRIPTION:
A stroke is a sudden loss of brain function. The interruption of blood flow or the rupture of blood vessels causes brain cells (neurons) in the affected area to die. The effects of a stroke depend on where the brain was injured, as well as how much damage occurred. A stroke can impact any number of areas including your ability to move, see, remember, speak, reason and read and write.

It is hereby postulated that irradiation using far infrared, with wavelength between 5 to 20 microns, of the central nervous system, the endocrine system and the whole body could prevent, control, manage or possibly lead to complete rehabilitation of people with stroke.

ELIGIBILITY:
Inclusion Criteria:

* People with Stroke

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Management and Cure of Stroke | 2 Years

SECONDARY OUTCOMES:
Rehabilitation of the following: ability to move, see, remember, speak, reason and read and write. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Principal Investigator — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada